CLINICAL TRIAL: NCT05199701
Title: Prospective Case Collection Study for New Mammography Technologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-08
Record Dates: First submitted 2021-12-16; First posted 2022-01-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Mammography
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Investigational Mammogram Exam (Experimental)
  Interventions: Device: Mammography

INTERVENTIONS:
Device: Mammography — All subjects who are indicated for a screening or diagnostic mammogram or breast biopsy will undergo an investigational exam in a new mammography device.

SUMMARY:
To evaluate the safety and efficacy of the proposed investigational device and assess its clinical utility in breast cancer screening and diagnosis to support continuing technology development of the investigational technology.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity.
* Subject is at least 35 years old.
* Subject is indicated for a screening or diagnostic mammogram or breast biopsy.

Exclusion Criteria:

* Subject is pregnant or thinks she may be pregnant
* Subject has breast implants, cardiac pacemakers, nipple piercings, or IV ports in the mammography field of view.
* Subject previously participated in the study.

Ages: 35 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinically acceptable image quality of the Investigational Device. | 4 years
  Questionnaire will be used to measure outcomes
Mammograms can be safety acquired on the Investigational Device. | 4 years
  Will be determined using the AE assessment.

SECONDARY OUTCOMES:
The ease of positioning and usability of the Investigational Device. | 4 years
  Questionnaire will be used to measure outcomes
Subject assessment of comfort of the Investigational Device. | 4 years
  Questionnaire will be used to measure outcomes

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Southwest Medical Imaging, Gilbert, Arizona
  - Scottsdale Medical Imaging LTD, Scottsdale, Arizona
  - Miami Breast Institute, Coral Gables, Florida
  - Diagnostic Centers of America Palm Beach Gardens, Palm Beach Gardens, Florida
  - Diagnostic Centers of America West Palm Beach, West Palm Beach, Florida
  - Baptist Health, Louisville, Kentucky
  - Progressive Radiology, Bel Air, Maryland
  - Corewell Health, Grand Rapids, Michigan
  - Elizabeth Wendy Breast Care, Rochester, New York
  - Solis Mammography Greensboro, Greensboro, North Carolina
  - Solis Mammography Columbus, Columbus, Ohio
  - Solis Mammography Burleson, Burleson, Texas
  - Washington Radiology, Arlington, Virginia
  - Washington Radiology, Sterling, Virginia

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and comply with the IRB. The IRB did not approved the secondary use of IPD at the time the protocol was approved.